CLINICAL TRIAL: NCT07395999
Title: Effectiveness of Pain Management Interventions in Patients With Chronic Cancer Pain in a Tertiary Care Hospital: A Retrospective Audit
Brief Title: Effectiveness of Pain Management Interventions in Patients With Chronic Cancer Pain
Status: Completed | Type: Observational
Sponsor: Aga Khan University (Other)
Responsible Party: Principal Investigator, Ali Sarfraz Siddiqui, Associate Professor, Aga Khan University
Other Study IDs: 2025-12152-38344
Record Dates: First submitted 2026-02-02; First posted 2026-02-09 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Chronic Cancer Pain; Pain Management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Chronic cancer pain: Patients with chronic cancer pain receiving pain management intervention
  Interventions: Other: Pharmacological and pain Intervention procedure

INTERVENTIONS:
Other: Pharmacological and pain Intervention procedure — Pain interventions ranges from pharmacological treatments including non-opioid analgesics, opioids and adjuvant analgesics to pain interventional procedures.

SUMMARY:
The goal of this observational study is to observe the effectiveness of pain management strategies in patients with chronic cancer pain presenting to pain management clinic at Aga Khan University.

The main question[s] it aims to answer are:

* What is the overall effectiveness of pain management techniques in patients with chronic cancer pain?
* What is the character and severity of pain?
* What is the frequency of pain intervention procedures?

ELIGIBILITY:
Inclusion Criteria:

* All adult patients
* Patients with chronic cancer pain

Exclusion Criteria:

* Patients lost to follow-up after the initial visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients presenting with chronic pain.
Sampling Method: Non-Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2025-11-14 (Actual); Primary Completion 2026-01-09 (Actual); Study Completion 2026-01-09 (Actual)

PRIMARY OUTCOMES:
Patient reported NRS score | Patient reported NRS score will be recorded at the first visit, and subsequent visit (till maximum three months) in the pain management clinic.
  Numeric Rating Score (NRS) is an 11-point scale with scores ranging from 0 (no pain) to 10 (worst imaginable pain), with higher scores indicating greater pain severity and therefore a worse outcome.

SECONDARY OUTCOMES:
Character of chronic pain | First and the follow-up visit ( till maximum three months) to the pain management clinic.
  Patients will be asked to describe the character (quality) of the pain they are experiencing e.g., burning, sharp, pricking, electric-shock-like.
Frequency of pain intervention procedure | At the end of three months.
  Pain intervention procedures undertaken by pain specialists for diagnostic or therapeutic purposes for the management of cancer pain

CONTACTS AND LOCATIONS:
Locations (1):
- Aga Khan University, Karachi, Pakistan, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided